CLINICAL TRIAL: NCT05705999
Title: Strengthening Tourette Treatment OPtions Using TMS to Improve CBIT, a Double-blind, Randomized, Controlled Study
Acronym: STOP-TIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: University of Florida (Other); Tourette Association of America (Other)
Responsible Party: Principal Investigator, Jessica Frey, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2211680481
Record Dates: First submitted 2023-01-21; First posted 2023-01-31 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome; Comprehensive Behavioral Intervention for Tics; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Tourette Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): Patients receiving active rTMS
  Interventions: Device: transcranial magnetic stimulation
- Sham rTMS (Sham Comparator): Patients receiving sham rTMS
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — The neurostimulation protocol will include 1-Hz rTMS over the bilateral SMA at 110% RMT. The SMA will be identified as 4 cm anterior to the vertex (Cz in standard 10-20 EEG setup). Each session will consist of 6 trains lasting 5 minutes each (300 pulses per train) with an intertrain interval of 1 minute for a total duration of 35 minutes (1800 pulses). Patients will receive 4 sessions each day on 4 consecutive days for a total of 16 sessions. Daily duration of this study protocol should last approximately 170 minutes including a 10-minute break in between each session

SUMMARY:
This pilot study will investigate the clinical and neurophysiological effects of repetitive transcranial magnetic stimulation (rTMS) followed by comprehensive behavioral intervention for tics (CBIT) in adult patients with Tourette's Syndrome (TS). Two groups of moderate disease severity will be randomized to receive active or sham rTMS targeted to the supplementary motor area (SMA) followed by eight CBIT sessions. The change in tic frequency and severity (primary outcome) and neurophysiological changes (secondary outcome) will be compared between the two groups. The central hypothesis is that low frequency rTMS will augment the effects of CBIT through favorable priming of the SMA network.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of Tourette Syndrome
* Moderate Tic Severity at baseline

Exclusion Criteria:

* Presence of metallic objects or neurostimulators in the brain
* Pregnancy
* History of active seizures or epilepsy
* Contraindications to receiving fMRI
* Inability to participate in CBIT due to other underlying cognitive or medical condition

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Through study completion, an average of 3 months
  Tic severity will be measured with YGTSS. YGTSS is a clinician-rated scale used to assess tic severity, scored out of 100 where a higher score indicates greater tic frequency and severity. It includes a checklist of motor and vocal tics followed by an assessment of the number, frequency, intensity, complexity, and inference of motor tics and phonic tics - scored separately. Each of these dimensions is scored on a 0 to 5 scale. The YGTSS provides three tic severity scores: Total Motor (0 to 25); Total Phonic (0 to 25) and the combined Total Tic Severity Score (0 to 50), as well as a separate Impairment dimension scored from 0 to 50.
Modified Rush Videotape Tic Rating Scale (mRVTRS) | Through study completion, an average of 3 months
  This is a tool used by an objective examiner to quantify the severity of a patient's tics by rating the number of body areas affected, motor tic frequency, phonic tic frequency, motor tic severity, and phonic tic severity, each on a 0 through 4 score by watching a video of the patient. Scored out of 20, where a higher score indicates greater tic severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Frey, MD, Principal Investigator — WVU RNI
Locations (1):
- WVU RNI, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No